CLINICAL TRIAL: NCT00610701
Title: Lateral Versus Anterior Spanning External Fixator for Tibial Plateau Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Extremely low enrollment and very little follow-up for meaningful data
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Crist, Associate Professor, Co-Director of Trauma Services, Co-Director of Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 1059937
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Fractures, Closed
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior pin placement (Experimental): Anterior pin placement
  Interventions: Device: Anterior pin placement
- Lateral pin placement (Experimental): Lateral pin placement
  Interventions: Device: Lateral pin placement

INTERVENTIONS:
Device: Anterior pin placement — Anteriorly-placed (front of the leg) femoral external fixator pins
  Arms: Anterior pin placement
Device: Lateral pin placement — Laterally-placed (side of the leg) femoral external fixator pind
  Arms: Lateral pin placement

SUMMARY:
The purpose of this study is to evaluate patients with tibial plateau fractures.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patients with tibial plateau fractures. The goal is to compare the differences between anteriorly placed (front of leg) femoral external fixator pins and laterally placed (side of leg) femoral external fixator pins.

Specifically, we are evaluating how this placement affects the quadriceps muscle and knee function. The parameters that will be assessed are knee function, pain, and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above (adult population)
* All open and closed tibial plateau fractures

Exclusion Criteria:

* 17 years of age and less (pediatric population)
* Quadriplegic patients
* Vascular Injury to Extremity
* Ipsilateral femur fractures
* Ipsilateral Hip fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-03; Primary Completion 2012-08 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Anterior: Anterior
  Anterior pin placement: Anteriorly-placed (front of the leg) femoral external fixator pins
- 2 Lateral: Lateral
  Lateral pin placement: Laterally-placed (side of the leg) femoral external fixator pind
Period: Overall Study
Arm/Group | 1 Anterior | 2 Lateral
Started | 15 | 20
Completed | 5 | 9
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Population: initially based on power analysis for anticipated quad strength data, final numbers based on those completing study in each group
Groups:
- 1-anterior Pin Placement: Anterior
  Anterior pin placement: Anteriorly-placed (front of the leg) femoral external fixator pins
- 2-lateral Pin Placement: Lateral
  Lateral pin placement: Laterally-placed (side of the leg) femoral external fixator pind
- Total: Total of all reporting groups
Arm/Group | 1-anterior Pin Placement | 2-lateral Pin Placement | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Strength
Description: measurement of quadriceps muscle strength at final followup = 1 year data at interim time points recorded, but only final reported for this purpose
Time Frame: (admission, 6 weeks, 3 months, 6 months) 1 year
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | 1-anterior Pin Placement | 2-lateral Pin Placement
Number analyzed (Participants) | 5 | 9
Nm | 35.9 (10.7) | 39.6 (17.7)
Statistical Analysis 1: Comparison: 1-anterior Pin Placement vs 2-lateral Pin Placement; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 year
Description: 14 patients completed the study
Arm/Group | 1 Anterior | 2 Lateral
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Anterior (N=5) | 2 Lateral (N=9)
death (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
infection (Infections and infestations) | 0 (0) | 1 (1) — knee infection
arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — knee arthrofibrosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No